CLINICAL TRIAL: NCT02683330
Title: Mindfulness-based Intervention for People Affected by Parkinson's Disease: A Distant-delivered Randomised Pilot Trial
Brief Title: Distant Delivery of a Mindfulness-based Intervention for People Affected by Parkinson's Disease
Acronym: MindPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: City, University of London (Other)
Responsible Party: Principal Investigator, Angeliki Bogosian, Lecturer in Psychology, City, University of London
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PSYETH (S/F) 15/16 112; Innovation grant: K-1409 (Other Grant/Funding Number: Parkinson's UK)
Record Dates: First submitted 2016-02-08; First posted 2016-02-17 (Estimated); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Parkinson's Disease
Keywords: PD; Parkinson's
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mindfulness-based intervention (MBI) (Experimental): Participants randomly assigned to the MBI group will receive 8 sessions over an 8-week period. The sessions will last 1 hour and will be held via video-conference through Skype, an online application.
  Interventions: Behavioral: Mindfulness-based intervention (MBI)
- Wait-list control (WLC) (No Intervention): Participants randomly assigned to the WLC group will be discouraged from any new mindfulness related activities during the trial. The WLC group will be offered the opportunity to take part in the MBI at the end of the 20-week follow-up.

INTERVENTIONS:
Behavioral: Mindfulness-based intervention (MBI) — MBI consists of 8 sessions and will cover becoming aware of emotions, thoughts and physical sensations, decentering and acceptance. Recordings of the body scan, a sitting meditation and a mindful movement meditation will be provided for daily home practice. Special care will be taken to address safety in the context of PD, and to adapt meditations to the physical limitations of PD.
  Arms: Mindfulness-based intervention (MBI)

SUMMARY:
Psychological difficulties, especially depression and anxiety are the most prevalent non-motor symptoms in Parkinson's Disease (PD). Pharmacological treatments are not as effective in PD. Mindfulness courses have received increased popularity and recognition as an effective way to manage emotional states, and there is ever growing findings of the effectiveness of mindfulness courses for people with long-term medical conditions. Two small pilot studies have indicated that mindfulness courses can be helpful for people with PD in improving symptoms of depression, language functioning and motor symptoms. The investigators propose to deliver these courses remotely, through Skype video conferences, to make it more accessible for people with mobility limitations and people who live in rural areas.

DETAILED DESCRIPTION:
This study will employ a mixed-methods design, with an experimental randomised control trial followed by a qualitative design. Sixty participants will be randomly assigned to the 8-week mindfulness course (n=30) or a wait-list control group (n=30). Block randomisation will be used and the randomisation scheme will be generated using the randomisation.com website. One-hour sessions will be delivered to groups of 5 people using Skype video-conferencing. As this is a pilot study analyses will largely be descriptive. Further, inferential analyses using mixed modelling will be conducted by intention-to-treat. At the end of the intervention, the investigators will interview the participants of the mindfulness group about their experiences of the course.

ELIGIBILITY:
Inclusion Criteria:

* be diagnosed with PD according to PD Brain Bank criteria by a neurologist or geriatrician
* have a computer and internet access at home, since the course will be delivered via Skype
* be able to communicate in English fluently
* be stabilised on mood altering medication and/or Parkinson's medication for a month

Exclusion Criteria:

* have severe cognitive impairment that would make participation in the mindfulness sessions and home practice of mindful meditation problematic or distressing. This will be assessed using the Telephone Interview for Cognitive Status-Modified (TICS-M, Brandt et al., 1993).
* have severe psychiatric conditions (e.g. psychosis, drug/ alcohol addiction) that can potentially risk failure in the treatment or limit participation in the course
* have severe hearing impairment
* are currently participating in other psychological therapies
* have prior formal training in mindfulness methods or current meditation practice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline Hospital Anxiety and Depression Scale (HADS) at 4, 8 and 20 weeks | Baseline, Mid-intervention (week 4), Post-intervention (week 8) and Follow-up (week 20).
  HADS also assessed at Mid-intervention (week 4), Post-intervention (week 8) and Follow-up (week 20) time points.

SECONDARY OUTCOMES:
Parkinson's Disease Activities of Daily Living Scale (PADLS) | Baseline, Mid-intervention (week 4), Post-intervention (week 8) and Follow-up (week 20)
Brief Pain Inventory (BPI) | Baseline, Mid-intervention (week 4), Post-intervention (week 8) and Follow-up (week 20)
Fatigue Severity Scale (FSS) | Baseline, Mid-intervention (week 4), Post-intervention (week 8) and Follow-up (week 20)
Insomnia Severity Index (ISI) | Baseline, Mid-intervention (week 4), Post-intervention (week 8) and Follow-up (week 20)

OTHER OUTCOMES:
Self-Compassion Scale (SCS) | Baseline, Mid-intervention (week 4), Post-intervention (week 8) and Follow-up (week 20)
Philadelphia Mindfulness Scale (PHLMS) | Baseline, Mid-intervention (week 4), Post-intervention (week 8) and Follow-up (week 20)
Experiences Questionnaire (EQ) | Baseline, Mid-intervention (week 4), Post-intervention (week 8) and Follow-up (week 20)
Acceptance Action Questionnaire (AAQ-II) | Baseline, Mid-intervention (week 4), Post-intervention (week 8) and Follow-up (week 20)
Subjective Well-Being questionnaire (SWB) | Baseline, Post-intervention (week 8) and Follow-up (week 20)
EuroQol Five-Dimensional questionnaire (EQ-5D-3L) | Baseline, Post-intervention (week 8) and Follow-up (week 20)
Visual Analogue Scale (VAS) | Baseline, Post-intervention (week 8) and Follow-up (week 20)
ICEpop CAPability measure for Adults (ICECAP-A) | Baseline, Post-intervention (week 8) and Follow-up (week 20)
Adult Social Care Outcomes Toolkit (ASCOT) | Baseline, Post-intervention (week 8) and Follow-up (week 20)

CONTACTS AND LOCATIONS:
Overall Officials: Angeliki Bogosian, PhD, Principal Investigator — City, University of London
Locations (1):
- City University London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pickut B, Vanneste S, Hirsch MA, Van Hecke W, Kerckhofs E, Marien P, Parizel PM, Crosiers D, Cras P. Mindfulness Training among Individuals with Parkinson's Disease: Neurobehavioral Effects. Parkinsons Dis. 2015;2015:816404. doi: 10.1155/2015/816404. Epub 2015 May 26. PMID 26101690
- [Background] Brandt J, Welsh KA, Breitner JC, Folstein MF, Helms M, Christian JC. Hereditary influences on cognitive functioning in older men. A study of 4000 twin pairs. Arch Neurol. 1993 Jun;50(6):599-603. doi: 10.1001/archneur.1993.00540060039014. PMID 8503796
- [Background] Cash, T. V., et al. (2015). Pilot Study of a Mindfulness-Based Group Intervention for Individuals with Parkinson's Disease and Their Caregivers. Mindfulness 1-11.
- [Derived] Bogosian A, Hurt CS, Vasconcelos E Sa D, Hindle JV, McCracken L, Cubi-Molla P. Distant delivery of a mindfulness-based intervention for people with Parkinson's disease: the study protocol of a randomised pilot trial. Pilot Feasibility Stud. 2017 Jan 16;3:4. doi: 10.1186/s40814-016-0117-4. eCollection 2017. PMID 28116120